CLINICAL TRIAL: NCT06098677
Title: Effect of Carotenoids Supplementation on Visual Function in Chinese Subjects Free of Retinal Disease: A Randomized Clinical Trial
Brief Title: Effect of Carotenoids Supplementation on Visual Function in Chinese Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Blackmores (China) CO., Ltd (Unknown)
Responsible Party: Principal Investigator, Xiaotong Han, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022KYPJ141
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotenoids group (Experimental): Participants in the intervention group receive oral supplementation of 10 mg L, 10 mg MZ and 2mg Z in a formula base oil suspension as one soft gel capsule in the morning per day. Each capsule contains 22 mg of carotenoids (10+10+2mg), thus each participant in the intervention group will receive a total of 22 mg of carotenoids per day.
  Interventions: Dietary Supplement: Carotenoids supplementation
- Placebo group (Placebo Comparator): Participants in the control group receive one soft gel capsule of placebo oil per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carotenoids supplementation — Daily oral supplementation of a soft gel capsule containing 10mg lutein (L), 10mg meso-zeaxanthin (MZ) and 2mg zeaxanthin (Z).
  Arms: Carotenoids group
Dietary Supplement: Placebo — Daily oral supplementation of a soft gel capsule containing only placebo oil
  Arms: Placebo group

SUMMARY:
The macula is a pigmented area at the center of the retina, and responsible for the central, high-resolution color vision. Age-related macular degeneration (AMD) is a disease of the macula and is the leading cause of irreversible vision impairment and blindness worldwide. The yellow pigment at the macula is referred to as macular pigment. There is now strong evidence showing that macular pigment (MP), which is composed of the dietary carotenoids lutein (L), meso-zeaxanthin (MZ), and zeaxanthin (Z) is protective against AMD and vision loss. MP is a powerful antioxidant and also filters short-wavelength (blue) light at the macula. The AREDS2 study concluded that supplementation of L and Z is beneficial for patients with non-advanced age-related macular degeneration (AMD). The CREST and other studies had reported that dietary supplementation of these carotenoids could enhance contrast sensitivity among the Caucasian population, whereas little information is known about the effect of dietary supplementation of carotenoids on contrast sensitivity among Chinese. Thus in this study, we aim to investigate whether supplementation of a formulation containing 10 mg L, 10 mg MZ, and 2mg Z on contrast sensitivity in Chinese subjects free of retinal disease. This study is a single-center, double-blinded, placebo-controlled, randomized clinical trial conducted at Zhongshan Ophthalmic Center (ZOC), Sun Yat-sen University, Guangzhou, China. Participants in the intervention group received oral supplementation of 10 mg L, 10 mg MZ, and 2mg Z in a formula base oil suspension as one soft gel capsule in the morning per day. Participants in the control group receive one soft gel capsule of placebo oil per day. The intervention and placebo supplements are identical in external appearance, and the two treatments are therefore indistinguishable from each other. The duration of the study intervention is 12 months, and study visits are conducted at baseline, 3 months, 6 months, and 12 months. The primary outcome measure is the change in contrast sensitivity (CS) at 6 cycles per degree (cpd) over the study course: Y=CS4-CS1, where CS1 is CS at 6 cpd at baseline, CS4 is the CS at 6cpd at the 12-month follow-up. The secondary outcomes of this study include CS at other cpds and at other study visits, best-corrected visual acuity, subjective visual function, and skin carotenoid levels at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects
* Age 35 years or above
* Monocular BCVA of 6/6 or better
* No more than +/- 5 diopters spherical equivalence of refraction
* No previous consumption of supplements containing macular carotenoids (L, Z and/or MZ) within the last 12 months
* Without severe retinal diseases (eg. retinal detachment, glaucoma, macular hole, idiopathic epiretinal membrane, retinitis pigmentosa, and age-related macular degeneration (assessed by experienced ophthalmologists during ocular examination)

Exclusion Criteria:

* Unable to provide informed consent
* With diagnosed diabetes
* With severe systemic disease which affects physical mobility and successful follow-up
* Contrast sensitivity at a spatial density of 6 cpd ≤ 1.5 % at baseline in the eye with better visual acuity
* Subjects who plan to receive cataract surgery within the next year
* Subjects who are unable to cooperate with the examinations during follow-ups, such as those who suffer from other serious systemic diseases or mental abnormalities
* History of intraocular surgery (eg. cataract surgery, vitrectomy and retinal laser photocoagulation)

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in contrast sensitivity (CS) at 6 cycles per degree (cpd) over 1 year | 1 year
  CS at 6 cpd at the 12-month follow-up minus CS at 6 cpd at baseline.

SECONDARY OUTCOMES:
CS at other cpds and at other study visits | 1 year
  CS at 1.2, 2.4, 9.6 and 15.15 cpd at baseline, 3-month follow-up, 6-month follow-up and 12-month follow-up; as well as CS at 6 cpd at 3-month follow-up and 6-month follow-up
Best-corrected visual acuity | 1 year
  Best-corrected visual acuity at baseline, 3-month follow-up, 6-month follow-up and 12-month follow-up
Subjective visual function | 1 year
  Subjective visual function measured by questionnaire at baseline, 3-month follow-up, 6-month follow-up and 12-month follow-up
Skin carotenoids score | 1 year
  Skin carotenoids score at baseline, 3-month follow-up, 6-month follow-up and 12-month follow-up

IPD SHARING:
Plan to Share IPD: No